CLINICAL TRIAL: NCT06185140
Title: Effects of Rehabilitation Programme on Respiratory Function in Patients with Acquired and Intervened Congenital Heart Disease: a Randomized Controlled Trial
Brief Title: Effects of Rehabilitation Programme on Respiratory Function in Patients with Acquired and Intervened Congenital Heart Disease.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Juan Luis Sanchez Gonzalez, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CardiorrespiUSAL
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Heart Defects, Congenital
Keywords: Exercise; Physiotherapy
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity

STUDY DESIGN:
Intervention Model Description: parallel randomized controlled trial with a simply assignment (1:1)
Who Masked: Outcomes Assessor
Masking Description: The study evaluator will not know the assignment of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Cardiac rehabilitation program
  Interventions: Other: cardiac rehabilitation program
- Control group (Active Comparator): These patients will complete the program from their home through the TELEA platform that belongs to SERGAS. They go to the hospital once at the beginning of the program to learn the program with the Physiotherapist and once again after a month. The program will be carried out twice a week for their home. Patients will be monitored during physical exercise with Garmin® heart rate monitors. Patients will download heart rate and Borg scale data after each session and can establish contact through the TELEA platform with the nursing staff of the Cardiac RHB Unit at all times.
  Interventions: Other: TELEA platform

INTERVENTIONS:
Other: cardiac rehabilitation program — Cardiac rehabilitation program
  Arms: Intervention group
Other: TELEA platform — TELEA platform
  Arms: Control group

SUMMARY:
Congenital heart defects (CHDs) are heart malformations that occur before birth, and they represent one of the leading causes of neonatal morbidity and mortality. they occur in approximately 1% of newborns and are associated with high morbidity and mortality rates. The etiology of these cardiac anomalies is mostly unknown. around 70-80% of cases are generated by the involvement of multiple affected genes combined with an environmental trigger that, when acting on a susceptible individual, promotes the expression of the damaged genome. maternal diseases during pregnancy or exposure to teratogenic substances are also implicated in the etiology.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with a history of cardiac transplantation or acquired congenital heart disease who have undergone at least one interventional procedure or surgical intervention at least 6 months before the start of the program in a state of clinical stability, hemodynamic stability, and ECG stability. They should have residual hemodynamic defects of sufficient severity that potentially restrict participation, and their perception of fragility may be influenced by the social, family, school environment, or by the patient themselves.
* Children aged 6-15 years at the start of the study.
* Children with maximum predicted oxygen consumption (VO2 max) values <80%, as measured in ergospirometry 6 months before the start of the intervention program.
* Patients for whom consultation with a pediatric cardiology specialist and pediatric rehabilitation specialist has not revealed contraindications for exercise.
* Children and their legal representatives should have provided informed consent and the ability to travel to the hospital center for in-person intervention.

Exclusion Criteria:

* Patients with acute, inflammatory, or infectious health conditions that could pose a risk to them during the course of the program.
* Patients who have undergone at least one interventional procedure or surgical intervention within a period of less than 6 months before the start of the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of respiratory function/spirometry | Baseline and immediately after the intervention
  Spirometry is the study of choice in pulmonary function laboratories. The parameters it measures are the volume of air that the child breathes in or out in absolute value or related to time, and is shown in the volume/time curve. The most useful functional parameters obtained after spirometry are forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), PEF and the FEV1 /FVC ratio

SECONDARY OUTCOMES:
Assessment of the respiratory musculature | Baseline and immediately after the intervention
  Volumetric Incentivator: The child will be placed in a seated position with feet on the floor and keeping the device in an upright position. The physiotherapist will ask the patient to exhale slowly and prolonged until the RV is reached and then perform a maximum inspiration through the mouthpiece ensuring lip sealing. The highest value of three procedures performed will be recorded as a reference for the intervention.
Functional capacity | Baseline and immediately after the intervention
  Pediatric treadmill ergospirometry will be used. This test is able to noninvasively evaluate the functional capacity of the child and to a lesser extent for the diagnosis of ischemic events

IPD SHARING:
Plan to Share IPD: No